CLINICAL TRIAL: NCT04533269
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study of Arnica Montana and Ledum Palustre Formulation on Mechanically Induced Bruising in Healthy Normal Volunteers
Brief Title: A Study of Topical Arnica & Ledum on Bruise Reduction in HNV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cearna, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CI-B001
Record Dates: First submitted 2020-08-24; First posted 2020-08-31 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-11

CONDITIONS: Bruise, Contusion
MeSH Terms: conditions — Contusions | interventions — Arnicae flos extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment kits will be coded. An unblinded statistician will provide the treatment codes after the study database is locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Arnica montana and Ledum palustre infused Pad
  Interventions: Other: Arnica montana, Ledum palustre
- Placebo (Placebo Comparator): Pad (Matching appearance with Active)
  Interventions: Other: Arnica montana, Ledum palustre

INTERVENTIONS:
Other: Arnica montana, Ledum palustre — Homeopathic

SUMMARY:
Subjects will have a bruise induced. A pad containing either a placebo or active will be applied to the bruise. Photographs will be taken over the following days to record bruise healing.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, crossover, multicenter study that will be used to evaluate the difference in bruise reduction efficacy between active remedy and placebo when a mechanical bruise is induced. The trial will be conducted at 5-8 sites with up to 150 subjects. Each subject will be injured two times using the same bruise-inducing mechanism, and the resulting bruises will be treated with active remedy or placebo-infused pads that will be identical in appearance. Subjects and study investigators will be blinded to the order of treatment assignment. Subjects will be asked to come to the clinic for photographic assessments of the bruise. Each subject will be randomly assigned to have a placebo or active remedy pad applied over each mechanically induced bruise on Day 1. The pad will be applied by study staff immediately after bruise induction (within 5 minutes). The pad will cover the bruised area completely, and then sealed with Tegaderm. All procedures, including bruise induction, treatment, and photography, will be administered by study staff who are blinded to treatment type. All photographs will be rated according to standardized criteria by blinded, trained study investigators after the completion of all subject data collection.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type 1-3
* BMI 25 kg/m2
* Self described bruisers
* Intact skin in the target area, free of markings, blemishes and hair

Exclusion Criteria:

* Use of recreational drugs, steroids, pain medications, other homeopathic remedies, anticoagulant therapies, antiplatelet therapy
* Known history of dermal sensitivity, serious illness, hematological abnormality, impaired wound healing
* Inability to forego application of topical products in the target area
* Hair removal by laser, wax or chemicals within one week prior to Day 1
* Avoid tanning beds
* History of allergy to topical gels, Arnica or Ledum
* Active wound or infection in the target area
* History of keloids or hypertrophic scarring
* History of collagen or vascular disease
* History of organ transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 11 days
  Time to bruise healing in active vs. placebo

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared and published.